CLINICAL TRIAL: NCT05432388
Title: A One Month, Investigator and Participant Blinded Study to Investigate the Efficacy and Safety of Remibrutinib (LOU064) at Multiple Dose Levels in Adult Participants With Peanut Allergy
Brief Title: Study of Efficacy, Safety and Tolerability of Remibrutinib in Adult Participants With an Allergy to Peanuts
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CLOU064I12201; 2021-006950-30 (EudraCT Number)
Record Dates: First submitted 2022-05-31; First posted 2022-06-27 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2025-05

CONDITIONS: Allergy, Peanut
Keywords: Groundnut Hypersensitivity; Hypersensitivity, Peanut; Peanut Allergy; Food Allergy; Oral food challenge; IgE; Remibrutinib; BTKi
MeSH Terms: conditions — Peanut Hypersensitivity; Food Hypersensitivity | interventions — remibrutinib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- remibrutinib low dose (Experimental): remibrutinib oral tablet
  Interventions: Drug: remibrutinib
- remibrutinib medium dose (Experimental): remibrutinib oral tablet
  Interventions: Drug: remibrutinib
- remibrutinib high dose (Experimental): remibrutinib oral tablet
  Interventions: Drug: remibrutinib
- placebo 3 week / remibrutinib low dose 1 week (Experimental): placebo oral tablet/ remibrutinib oral tablet
  Interventions: Drug: remibrutinib; Drug: placebo
- placebo (Placebo Comparator): oral tablet
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: remibrutinib — oral tablets
  Other Names: (LOU064)
  Arms: placebo 3 week / remibrutinib low dose 1 week; remibrutinib high dose; remibrutinib low dose; remibrutinib medium dose
Drug: placebo — oral tablets
  Arms: placebo; placebo 3 week / remibrutinib low dose 1 week

SUMMARY:
A study to evaluate the safety, efficacy and tolerability of remibrutinib at three doses versus placebo in adult participants who have a confirmed allergy to peanuts. The efficacy will be measured by the ability of participants to tolerate increasing doses of peanut protein during an oral food challenge after 1 month of study treatment.

DETAILED DESCRIPTION:
This is a one month, phase 2, multi-center, randomized, investigator- and participant-blinded, placebo controlled study to assess the safety, efficacy and tolerability of remibrutinib (LOU064) in 3 doses of oral tablet twice a day in participants with a medically confirmed diagnosis of IgE-mediated peanut allergy. Participants will be randomized to remibrutinib low, medium or high dose for one-month treatment period (up to 5 weeks). Participants will have oral food challenges at the beginning of the study and at the end of the treatment period to assess their symptoms from increasing doses of peanut allergen.

ELIGIBILITY:
Inclusion Criteria:

* Medical History of allergy to peanuts
* Positive peanut IgE >= 0.35 kUA/L
* Positive Skin Prick test for peanut allergen during screening for study
* Positive Oral Food Challenge to peanut during screening for study
* Willingness to comply with study schedule and procedures and avoid other allergens during study period

Exclusion Criteria:

* History of severe or life-threatening hypersensitivity event leading to ICU admission or intubation within 60 days of screening
* Uncontrolled asthma
* Bleeding risk or coagulation disorder(s)
* Use of anticoagulants or anti-platelets (aspirin or clopidogrel may be permitted)
* History of splenectomy
* Any significant disease that would put the safety of the patient at risk. This includes, but is not limited to: history of cancer, significant cardiac disease/history, hematology disorders, history of GI bleeding, active infectious process, liver disease, renal disease, immunologic disease (stable diabetes and thyroid disease may be permitted), alcohol or drug abuse, etc.

Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 76 (Actual)
Dates: Start 2022-10-12 (Actual); Primary Completion 2025-03-11 (Actual); Study Completion 2025-03-11 (Actual)

PRIMARY OUTCOMES:
Efficacy or oral remibrutinib compared to placebo, as measured by the proportion of participants who can tolerate a single dose of >=600mg of peanut protein without dose-limiting symptoms during DBPCFC | Baseline and Day 26
  Responder status defined as tolerating a single dose of >=600mg of peanut protein without dose-limiting symptoms during the DBPCFC

SECONDARY OUTCOMES:
Efficacy or oral remibrutinib compared to placebo, as measured by the proportion of participants who can tolerate a single dose of >=1000mg of peanut protein without dose-limiting symptoms during DBPCFC | Baseline, Days 26 and 28
  Responder status defined as tolerating a single dose of >=1000mg of peanut protein without dose-limiting symptoms during the DBPCFC
Efficacy or oral remibrutinib compared to placebo, as measured by the proportion of participants who can tolerate a single dose of >=3000mg of peanut protein without dose-limiting symptoms during DBPCFC | Baseline, Days 26 and 28
  Responder status defined as tolerating a single dose of >=3000mg of peanut protein without dose-limiting symptoms during the DBPCFC
Efficacy or oral remibrutinib compared to placebo as measured by the madimum symptoms severity at any single challenged dose up to and including 1000mg of peanut protein | Baseline, Days 26 and 28
  Maximum severity of symptoms occurring at any challenge dose of peanut protein up to and including 1000mg during the DBPCFC
Efficacy of 3 weeks placebo treatment followed by 1 week of oral remibrutinib treatment compared to placebo as measured by the proportion of participants who can tolerate a single dose of >=600mg peanut protein during DBPCFC | Baseline, Days 26 and 28
  Responder status defined as tolerating a single dose of >=600mg peanut protein without dose limiting symptoms during the DBPCFC
Effects of multiple doses of remibrutinib compared to placebo, as measured by multiple systemic biomarkers to inform on response to treatment or disease severity | Baseline, Days 26 and 28
  Change from baseline at weeks 1 and 4 of peanut specific IgE and IgG4, including peanut components
Ability of remibrutinib to impact skin mast cells through the assessment of allergen-specific skin prick test | Baseline and Day 26
  Change from screening in skin prick test wheal diameters
Cmax of remibrutinib | Day 8 and Day 25
  Remibrutinib concentrations in blood and PK parameter - Cmax
AUClast of remibrutinib | Day 8 and Day 25
  Remibrutinib concentrations in blood and PK parameter - AUClast
AUCtau of remibrutinib | Day 8 and Day 25
  Remibrutinib concentrations in blood and PK parameter - AUCtau
Tmax of remibrutinib | Day 8 and Day 25
  Remibrutinib concentrations in blood and PK parameter - Tmax

CONTACTS AND LOCATIONS:
Locations (23):
- United States (23):
  - Allervie Clinical Research, Birmingham, Alabama
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - California Allergy and Asthma Medical Group, Los Angeles, California
  - Allergy and Asthma Clin Res Inc, Walnut Creek, California
  - Asthma and Allergy Associates P C, Colorado Springs, Colorado
  - Colorado Allergy and Asthma Ctr PC, Denver, Colorado
  - Childrens National Hospital, Washington D.C., District of Columbia
  - Treasure Valley Medical Research, Boise, Idaho
  - Midwest Allergy Sinus Asthma SC, Normal, Illinois
  - Asthma and Allergy Center of Chicago S C, River Forest, Illinois
  - Bluegrass Allergy Research ., Lexington, Kentucky
  - Family Allergy and Asthma, Louisville, Kentucky
  - Johns Hopkins Hospital, Baltimore, Maryland
  - Institute for Asthma and Allergy PC, Chevy Chase, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - University of Michigan Clinical Trials Office, Ann Arbor, Michigan
  - CenExel HRI, Berlin, New Jersey
  - Columbia University Irving Medical, New York, New York
  - CR Services Acquisition US Main center, Columbus, Ohio
  - Vital Prospects Clinical Research Institute, Tulsa, Oklahoma
  - Western Sky Medical Research, El Paso, Texas
  - Allergy Associates of Utah, Sandy City, Utah
  - Seattle Allergy and Asthma Rsch, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com